CLINICAL TRIAL: NCT02427542
Title: A Brief Cognitive Behavioural Therapy (CBT) Intervention for Depersonalisation/Derealisation in Psychosis: a Feasibility Study
Brief Title: Feasibility Trial of CBT for Depersonalisation in Psychosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol 141216v3; 15/LO/0081 (Other: Research Ethics Committee); 166784 (Other: IRAS); R&D2015/017 (Other: R&D office)
Record Dates: First submitted 2015-04-08; First posted 2015-04-28 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-02

CONDITIONS: Psychotic Disorders; Depersonalization
Keywords: Randomized Controlled Trial
MeSH Terms: conditions — Psychotic Disorders; Depersonalization | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT for DP (Active Comparator): Six sessions of CBT covering psycho-education, formulation, enhancing coping strategies (including grounding) and cognitive restructuring techniques.
  Interventions: Other: CBT for Depersonalization/Derealization
- Treatment as usual (Placebo Comparator): Participants will continue to receive their normal treatment - in most cases, this will be care coordination/case management delivered through a community mental health team and may include medication.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: CBT for Depersonalization/Derealization — In addition to treatment as usual, six sessions of Cognitive Behavioural Therapy for Depersonalization/Derealisation covering psychoeducation, formulation, coping strategies.
  Arms: CBT for DP
Other: Treatment as usual — Treatment as usual - in most cases case management/care coordination and may include medication
  Arms: Treatment as usual

SUMMARY:
This is a feasibility trial designed to test the feasibility and acceptability of a brief form (six sessions) of Cognitive Behavioural Therapy (CBT) for Depersonalisation/Derealisation (DP/DR) in those individuals who also have a diagnosis of a psychotic disorder. Participants will be randomised to receive either six sessions of CBT targeting DP/DR symptoms or to a treatment as usual control condition.

DETAILED DESCRIPTION:
Depersonalisation/derealisation (DP/DR) are distressing symptoms of having a sense of detachment and unreality about oneself (DP) or the external world (DR). Cognitive Behavioural Therapy (CBT) has been found to be beneficial in treating patients with chronic DP/DR. CBT for DP/DR includes educating patients about these experiences so they have a better understanding and less fear; teaching ways of coping to help them manage the symptoms better; helping reduce the impact on their day to day functioning; and working together to find less distressing ways of interpreting these experiences. Recent research has highlighted that DP/DR symptoms are common in people diagnosed with psychotic disorders, and when present are linked with more severe psychotic symptoms. However, there has been no previous study to ascertain if CBT to target DP/DR in psychosis would be effective. This study therefore aims to establish the feasibility of a brief CBT intervention for DP/DR in people diagnosed with a psychotic disorder. It is hoped that the CBT will reduce the distress associated with DP/DR experiences, with a possibility of reducing psychotic phenomena in addition. The investigators will seek to recruit adults aged 18-70 with a current psychotic symptoms as well as meeting threshold for DP/DR disorder. Participants will be randomly assigned to receive six sessions of CBT or to a treatment as usual control. Outcomes will be assessed at baseline and follow-up interview at 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* current experience of psychotic symptoms,
* meeting threshold for DP/DR disorder (scores greater than 70 on Cambridge Depersonalization Scale (CDS)).

Exclusion Criteria:

* insufficient capacity to provide informed consent;
* insufficient proficiency in English (spoken and written) to engage in CBT;
* a primary diagnosis of intellectual disability, head injury, substance misuse or organic cause for psychosis;
* those currently engaging in CBT or other psychotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention ( including recruitment rates, acceptance rates, drop outs) | 10 weeks
  Feasibility estimates of delivering the intervention including recruitment rates, acceptance rates, drop outs.
Depersonalisation score (Score on the Cambridge Depersonalisation Scale) | 10 weeks
  Score on the Cambridge Depersonalisation Scale
Acceptability of intervention (Satisfaction and attrition rates) | 10 weeks
  Satisfaction and attrition rates

SECONDARY OUTCOMES:
Depression (Score on Beck Depression Inventory) | 10 weeks
  Score on Beck Depression Inventory
Anxiety (Score on Beck Anxiety Inventory) | 10 weeks
  Score on Beck Anxiety Inventory
Psychosis (Score on the Psychotic Symptom Rating Scale (PSYRATS) | 10 weeks
  Score on the Psychotic Symptom Rating Scale (PSYRATS)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Farrelly, PhD, Principal Investigator — King's College London
Locations (1):
- PICUP clinic, London, London, United Kingdom

REFERENCES:
- [Derived] Farrelly S, Peters E, Azis M, David AS, Hunter ECM. A brief CBT intervention for depersonalisation-derealisation disorder in psychosis: Results from a feasibility randomised controlled trial. J Behav Ther Exp Psychiatry. 2024 Mar;82:101911. doi: 10.1016/j.jbtep.2023.101911. Epub 2023 Sep 12. PMID 37716893
- [Derived] Farrelly S, Peters E, Azis M, David A, Hunter EC. A brief CBT intervention for depersonalisation/derealisation in psychosis: study protocol for a feasibility randomised controlled trial. Pilot Feasibility Stud. 2016 Aug 11;2:47. doi: 10.1186/s40814-016-0086-7. eCollection 2016. PMID 27965864